CLINICAL TRIAL: NCT05536037
Title: Metformin Chemoprevention of Oral Premalignant Lesions
Brief Title: Metformin for the Prevention of Oral Cancer in Patients With Oral Premalignant Lesions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22D.296; JT 17064 (Other: JeffTrial Number)
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Erythroplakia; Leukoplakia; Oral Cavity Carcinoma; Proliferative Verrucous Leukoplakia
MeSH Terms: conditions — Erythroplasia; Leukoplakia; Mouth Neoplasms | interventions — Metformin; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (metformin) (Experimental): Patients receive metformin PO QD on days 1-3 and then PO BID for up to 12 months in the absence of unacceptable toxicity.
  Interventions: Drug: Metformin; Procedure: Biopsy

INTERVENTIONS:
Drug: Metformin — Given PO
  Other Names: 1-Dimethylbiguanide; 657-24-9; N-dimethylbiguanide; N-Dimethylimidodicarbonimidic Diamide
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase I trial tests whether metformin works in reducing the annual transformation (development of invasive cancer) of oral precancerous lesions into cancerous lesions. Metformin is a drug approved for the treatment of diabetes, but studies have shown that it may have some anticancer properties. Giving metformin may help prevent or slow the development of oral cancer from precancerous lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the transformation-free-survival in lesion types erythroplakia (EP) and verrucous hyperplasia (VH). 'Transformation' is defined as the development of invasive cancer.

SECONDARY OBJECTIVE:

I. To evaluate the current spontaneous regression rates, i.e., percentages of patients having lesion disappear within 1-year post treatment, in all four lesion types and compare them with historical documented regression rate in literature.

EXPLORATORY OBJECTIVE:

I. To evaluate the transformation-free-survival in lesion types homogenous leukoplakia (HL) and non-homogenous leukoplakia (NHL).

OUTLINE:

Patients receive metformin orally (PO) once daily (QD) on days 1-3 and then PO twice daily (BID) for up to 12 months in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Clinical appearance of lesion

  * Homogenous leukoplakia
  * Non- homogenous leukoplakia
  * Erythroplakia
  * Proliferative verrucous leukoplakia
* Histologic appearance

  * No dysplasia
  * Mild dysplasia
  * Moderate dysplasia
  * Severe dysplasia
* Diabetics: if on metformin, will get them to 2000 mg per day, if not, will add metformin in consultation with endocrinologist
* All subjects must be able to comprehend and sign a written informed consent document
* Willing and able to be available for the duration of the study
* In general good health with no contraindication to biopsy or metformin therapy
* Laboratory results

Exclusion Criteria:

* Carcinoma in-situ, verrucous carcinoma, invasive squamous cell carcinoma (SCCa)
* Exclude systemic causes of the lesion: pemphigus, pemphigoid, systemic lupus erythematosus (SLE), lichenoid drug reaction, human immunodeficiency virus (HIV), syphilis
* Exclude local inciting factors: rule out (r/o) but allowing 2 weeks to pass and see if there is resolution, if not and doesn't resolve with local measures, medical treatment, enroll

  * Frictional: sharp tooth
  * Trauma
* Immunosuppression by natural illness or medically induced
* Hypersensitivity or allergic reaction to metformin or some other contraindication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Transformation-free-survival, in lesion types erythroplakia and verrucous hyperplasia | Up to 3 years
  Will be summarized using Kaplan-Meier curves as well as 95% confidence ands. Kaplan-Meier estimates of the 3-year transformation-free-survival rates will be reported with 95% confidence interval. One-sample two-sided log-rank test will be applied to all four lesions as well.

SECONDARY OUTCOMES:
Change in lesion status | Baseline to 1 year after treatment
  Evaluated on a Likert-scale with three levels: 'worsen', 'same' and 'disappear', compared to each patient's baseline lesion status (as measured at pre-treatment and one year post initiation of treatment). The lesion size and status evaluated at 1-year post-treatment will be summarized using percentages as well as 95% Clopper-Pearson exact confidence intervals. The current spontaneous regression rates (i.e., percentage of 'disappear') will be compared against the historically documented regression rate of 35% using two-sided exact binomial test.

OTHER OUTCOMES:
Transformation-free-survival, in lesion types homogenous leukoplakia and non-homogenous leukoplakia | Up to 3 years
  Will be summarized using Kaplan-Meier curves as well as 95% confidence ands. Kaplan-Meier estimates of the 3-year transformation-free-survival rates will be reported with 95% confidence interval. One-sample two-sided log-rank test will be applied to all four lesions as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States